CLINICAL TRIAL: NCT06699303
Title: Study of the Effect of Breast Milk and Hamamelis Virginiana (Potency12MG/100G) on the Healing of Diaper Dermatitis in Infants
Brief Title: Effect of Breast Milk on Diaper Dermatitis in Infants
Acronym: dermatit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E-16214662-050.01.04-220310-04
Record Dates: First submitted 2023-12-25; First posted 2024-11-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diaper Dermatitis
Keywords: diaper dermatitis; mother's milk; hamamelı̇s vı̇rgı̇nı̇nana
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Intervention Model Description: It was planned as a randomized controlled and single blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uncomplicated Diaper Dermatitis Severity Assessment Scale in Babies (Experimental): In the study, a data collection form consisting of 13 questions regarding the sociodemographic characteristics of 0-12 month old babies and the "Uncomplicated Diaper Dermatitis Severity Assessment Scale in Babies, developed by Buckley et al. in 2016 and whose Turkish validity and reliability studies were conducted by Keskin, will be used.
  Interventions: Other: Use of diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g / 100 g for infants in the control group in diaper dermatitis care

INTERVENTIONS:
Other: Use of diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g / 100 g for infants in the control group in diaper dermatitis care — In diaper dermatitis care, it was planned to use their mothers' milk for the babies in the experimental group and diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g/100g for the babies in the control group. The reason why diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g/100 g is preferred is that it is the most frequently used cream in cases of uncomplicated diaper dermatitis. The mothers of the babies in the control group will be asked to wash and dry the baby's diaper with soap and water during each diaper change and then apply diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g/100 g. Mothers will be asked to record any new signs and symptoms that develop during the treatment and to inform the investigators will be asked to provide information. Positive and negative effects of treatment will also be recorded.
  Other Names: Administration of mother's milk for infants in the experimental group in the care of diaper dermatitis

SUMMARY:
Diaper dermatitis, one of infants' most common health problems, can be treated with various methods. One of these methods is breast milk. Studies show that breast milk is a non-harmful, accessible and effective product in the healing of dermatitis. This study was planned to be a randomized, controlled, and single-blinded study to evaluate the effect of breast milk and diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g/100g on the healing process in 0-12-month-old infants with diaper dermatitis. The population of the study consisted of 0-12 months old infants with diaper dermatitis who applied to the Pediatrics Outpatient Clinic of X Hospital. Since not all infants with diaper dermatitis complaints were examined, the number of the population cannot be known. The sample size was calculated as 26 for each group and 52 in total . 30 infants were planned to be included in each group. The licensed IBM SPSS 22.0 (Statistical Package for the Social Sciences) package program will be used for statistical data analysis. Standard deviation, number and percentage will be used in data analysis. Man Whitney U test and Fisher exact test (repeated measures) will be used to evaluate whether there is a difference between independent groups. For the significance level of the data, 0.05 will be used.

DETAILED DESCRIPTION:
Diaper dermatitis, one of the most common health problems in infants, can be treated with various methods (Blume-Peytavi Kanti, 2018; Gozen et al., 2014; Seifi, Jalali, Heidari, 2017). One of these methods is breast milk. Breast milk has strong immunologic properties that protect infants from respiratory diseases, middle ear infections and gastrointestinal system diseases. It also has protective effects against diabetes mellitus, obesity, hyperlipidemia, hypertension, cardiovascular diseases, autoimmunity and asthma. Because of these positive properties, breast milk has lifelong positive effects. In recent years, studies on the effect of breast milk in the treatment of dermatitis have been increasing (Kasrae, Farahani, Yousefi, 2015, Blume-Peytavi Kanti, 2018; Gozen et al., 2014; Seifi, Jalali, Heidari, 2017, Bener et al., 2007). In a study conducted by Gozen et al. using breast milk and barrier cream, barrier cream was found to be more effective than breast milk, especially in the treatment of moderate and severe dermatitis (Gozen et al., 2014). Farahani et al. applied 1% hydrocortisol and breast milk for 7 days in a randomized controlled study on diaper dermatitis. In this study, improvement was found to be similar on the 3rd and 7th days of treatment and it was concluded that breast milk was safe and effective (Farahani, Ghobadzadeh, Yousefi, 2013) Seifi et al. found a statistically significant difference between the groups in favor of breast milk in terms of skin rash score on the first and third days of the application in their study using breast milk in diaper rash care (p=0.013, p=0.005, respectively). This difference was even more significant on the fifth day (p=0.004, p=0.001) (Seifi et al., 2017). Studies show that breast milk is a non-harmful, free and effective product for the healing of dermatitis.

This study was planned to be a randomized, controlled, and single-blinded study to evaluate the effect of breast milk and diaper rash cream containing Hamamelis virginiana (potency 12mg/100g) 5.35 g/100g on the healing process in 0-12-month-old infants with diaper dermatitis. The population of the study consisted of 0-12 months old infants with diaper dermatitis who applied to the Pediatrics Outpatient Clinic . Since not all infants with diaper dermatitis complaints were examined, the number of the population cannot be known. The sample size was calculated as 26 for each group and 52 in total with the "A priori. 30 infants were planned to be included in each group. The licensed IBM SPSS 22.0 (Statistical Package for the Social Sciences) package program will be used for statistical data analysis. Standard deviation, number and percentage will be used in data analysis. Man Whitney U test and Fisher exact test (repeated measures) will be used to evaluate whether there is a difference between independent groups. For the significance level of the data, 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Babies fed with breast milk,
* Healthy babies aged 0-6 months,
* Babies who do not have diarrhea or thrush at the time of application,
* Fungus, eczema, allergic disease, etc.Babies without a history of skin disease,
* Babies who do not use antimycotic drugs (Ampotericin etc.), antibiotics and steriods ---before and during the application,
* Babies who do not apply medication or other materials (barrier creams, powder and other medications) to the dermatitis area.

Exclusion Criteria:

* Babies who are not breastfed
* Those who did not agree to participate in the study

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
It will be evaluated whether there is a difference between breast milk and dermatitis cream in terms of healing diaper dermatitis in babies aged 0-12 months. | 6 months
  Data will be collected using the baby identification form and the Infant Uncomplicated Diaper Dermatitis Severity Rating Scale (UCDAS).

CONTACTS AND LOCATIONS:
Overall Officials: Döndü 1 Sevimli Güler, PhD, Principal Investigator — Sakarya Training and Research Hospital; Zekiye 4 Turan, PhD, Study Director — Sakarya University
Locations (2):
- Turkey (Türkiye) (2):
  - Sakarya Training and Research Hospital, Sakarya, Adapzarı
  - Sakarya Üniversitesi, Sakarya, Adapzarı

IPD SHARING:
Plan to Share IPD: No
Our study findings have not yet been published.